CLINICAL TRIAL: NCT05380687
Title: Time Course of Neuro-ventilatory Efficiency During a Spontaneous Breathing Training
Acronym: TONES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 002418
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2023-06

CONDITIONS: Ventilator Weaning; Respiration, Artificial; Respiratory Muscles; Respiratory Failure; Critical Care
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomized crossover of 2 trainings (A and B)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training A - PEEP 10-5-5-5 (Experimental): The respiratory muscles of all participants will be trained in 4 consecutive blocks of 30 minutes during ventilation in neural pressure support mode (NPS) with a pressure support of 7 cmH2O.
  During training A, the 4 blocks are
  A1. PEEP 10 cmH2O | A2. PEEP 5 cmH2O | A3. PEEP *5* cmH2O | A4. PEEP 5 cmH2O
  During the training, ventilator data will be recorded and respiratory muscles will be imaged using ultrasound.
  Before and after each training block, an inspiratory and an expiratory hold (both ≤ 30 seconds) will be performed to assess fatigue.
  Interventions: Diagnostic Test: Inspiratory hold; Diagnostic Test: Expiratory hold; Diagnostic Test: Ultrasound of respiratory muscles; Other: PEEP 10; Other: PEEP 5
- Training B - PEEP 10-5-0-5 (Experimental): The respiratory muscles of all participants will be trained in 4 consecutive blocks of 30 minutes during ventilation in neural pressure support mode (NPS) with a pressure support of 7 cmH2O.
  During training B, the 4 blocks are
  B1. PEEP 10 cmH2O | B2. PEEP 5 cmH2O | B3. PEEP *0* cmH2O | B4. PEEP 5 cmH2O
  During the training, ventilator data will be recorded and respiratory muscles will be imaged using ultrasound.
  Before and after each training block, an inspiratory and an expiratory hold (both ≤ 30 seconds) will be performed to assess fatigue.
  Interventions: Diagnostic Test: Inspiratory hold; Diagnostic Test: Expiratory hold; Diagnostic Test: Ultrasound of respiratory muscles; Other: PEEP 10; Other: PEEP 5; Other: PEEP 0

INTERVENTIONS:
Diagnostic Test: Inspiratory hold — A short period (< 30 seconds) during which both inspiratory and expiratory valves of the ventilator circuit are closed at the end of inspiration. It is used to asses expiratory force generation (maximal expiratory pressure, MEP) and frequently used in clinical practice.
Diagnostic Test: Expiratory hold — A short period (< 30 seconds) during which both inspiratory and expiratory valves of the ventilator circuit are closed at the end of expiration. It is used to asses static PEEP and inspiratory force generation (maximal inspiratory pressure, MIP & occlusion pressure, ∆Pocc) and is frequently used in clinical practice.
Diagnostic Test: Ultrasound of respiratory muscles — Ultrasound of the diaphragm, parasternal intercostal muscle and internal oblique muscle will be performed during each block. Thickening fractions, calculated as thickness at end-inspiration minus thickness at end-expiration divided by thickness at end-expiration, are used to assess the contribution of the muscle to the tidal volume. A median over 5 breaths will be calculated.
Other: PEEP 10 — Positive End-Expiratory Pressure of 10cmH2O for 30 minutes
Other: PEEP 5 — Positive End-Expiratory Pressure of 5cmH2O for 30 minutes
Other: PEEP 0 — Positive End-Expiratory Pressure of 0cmH2O for 30 minutes
  Arms: Training B - PEEP 10-5-0-5

SUMMARY:
The TONES trial aims to evaluate the neuroventilatory efficiency (NVE = tidal volume / peak voltage of diaphragm contraction) measured during a zero-assist manoeuvre (ZAM, i.e. with PEEP but without pressure support). This novel parameter, NVE-ZAM, will be studied in a blocked, crossover, repeated measures design.

Possible confounders, such as activity of respiratory muscles other than the diaphragm, are included.

The investigators hypothesized that

* the NVE during a zero-assist maneuver has a low variability and high repeatability at the same level of PEEP (within subjects, within blocks)
* NVE-ZAM trends differ between participants (between subjects, within blocks) and between PEEP levels (within subjects, between blocks)

The primary aim is to study the variability and repeatability of the NVE-ZAM within subjects and within blocks.

Additionally, the effect of PEEP, muscle fatigue and recruitment of the accessory and expiratory muscles of respiration on the NVE-ZAM will be studied in an exploratory analysis (in multiple combinations of within and between subjects and/or blocks).

ELIGIBILITY:
Inclusion criteria:

* adult (18-80 yrs.)
* admitted to the ICU
* intubated and mechanically ventilated
* Edi catheter (Maquet, Solna, Sweden) in situ as part of their clinical care
* ventilated in a support mode (e.g. pressure support) with a support between 7 and 15 cmH2O, a PEEP ≤10 cmH2O and an Fi02 <0.6, all since ≥6 hours.
* can participate in the trial as judged by their attending physician

Exclusion criteria:

* pregnancy
* refusal of participation
* pre-existing neuromuscular disorders (e.g., Guillain-Barré)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Neuroventilatory efficiency (NVE) during a zero-assist breath in neural pressure support mode with a pressure support level of 7cmH2O and a PEEP of 10 cmH2O | Measured each 3 mintues during blocks A1 and B1: initial 30 minutes of training in both trainings A and B (cumulative: 2x 30 minutes)
  Measured using an Edi catheter (Maquet, Solna, Sweden) each 3 minutes as tidal volume / delta Edi.
  Zero assist is defined as a pressure support of 0 cmH2O during a single breath.
Neuroventilatory efficiency (NVE) during a zero-assist breath in neural pressure support mode with a pressure support level of 7cmH2O and a PEEP of 5 cmH2O | Measured each 3 mintues during blocks A2 and B2: second next 30 minutes of training in both trainings A and B (cumulative: 2x 30 minutes)
  Measured using an Edi catheter (Maquet, Solna, Sweden) each 3 minutes as tidal volume / delta Edi.
  Zero assist is defined as a pressure support of 0 cmH2O during a single breath.
Neuroventilatory efficiency (NVE) during a zero-assist breath in neural pressure support mode with a pressure support level of 7cmH2O and a PEEP of 5 cmH2O | Measured each 3 mintues during block A3: third next 30 minutes of training in training A (cumulative: 1x 30 minutes)
  Measured using an Edi catheter (Maquet, Solna, Sweden) each 3 minutes as tidal volume / delta Edi.
  Zero assist is defined as a pressure support of 0 cmH2O during a single breath.
Neuroventilatory efficiency (NVE) during a zero-assist breath in neural pressure support mode with a pressure support level of 7cmH2O and a PEEP of 0 cmH2O | Measured each 3 mintues during block B3: third next 30 minutes of training in training B (cumulative: 1x 30 minutes)
  Measured using an Edi catheter (Maquet, Solna, Sweden) each 3 minutes as tidal volume / delta Edi.
  Zero assist is defined as a pressure support of 0 cmH2O during a single breath.
Neuroventilatory efficiency (NVE) during a zero-assist breath in neural pressure support mode with a pressure support level of 7cmH2O and a PEEP of 5 cmH2O | Measured each 3 mintues during blocks A4 and B4: fourth next 30 minutes of training in both trainings A and B (cumulative: 2x 30 minutes)
  Measured using an Edi catheter (Maquet, Solna, Sweden) each 3 minutes as tidal volume / delta Edi.
  Zero assist is defined as a pressure support of 0 cmH2O during a single breath.

SECONDARY OUTCOMES:
Change in RSBI (ml*min) | Measured at each breath during 30 minutes in block B3 (at zero PEEP; cumulative 30 minutes)
  Rapid shallow breathing index, calculated as tidal volume divided by respiratory rate
Change in P0.1 (cmH2O) | Measured at each breath during 30 minutes for each training block (A1-4 & B1-4; cumulative 4hours)
  Airway pressure at the first 100 milliseconds of a breath
Change in Cdyn (ml / cmH2O) | Measured at each breath during 30 minutes for each training block (A1-4 & B1-4; cumulative 4hours)
  Dynamic respiratory system compliance, calculated as tidal volume divided by driving pressure
Change in Raw (cmH2O * L / s) | Measured at each breath during 30 minutes for each training block (A1-4 & B1-4; cumulative 4hours)
  Respiratory system resistance, calculated as (peak inspiratory pressure - plateau pressure) / flow
Change in PIP (cmH2O) | Measured at each breath during 30 minutes for each training block (A1-4 & B1-4; cumulative 4hours)
  Peak Inspiratory Pressure
Change in DTF | Measured for 5 breaths in the 30 minutes for each training block (A1-4 & B1-4; cumulative 4hours)
  Diaphragm thickening fraction, calculated as (diaphragm thickness at end-inspiration - diaphragm thickness at end-expiration) / diaphragm thickness at end-expiration [dimensionless]. Muscle thickness will be measured in millimeters using M-mode ultrasound with the probe placed perpendicular to the muscle (not including the thickness of fascial muscle layers).
Change in ICTF | Measured for 5 breaths in the 30 minutes for each training block (A1-4 & B1-4; cumulative 4hours)
  Parasternal intercostal muscle thickening fraction, calculated as (parasternal intercostal muscle thickness at end-inspiration - parasternal intercostal muscle thickness at end-expiration) / parasternal intercostal muscle thickness at end-expiration [dimensionless]. Muscle thickness will be measured in millimeters using M-mode ultrasound with the probe placed perpendicular to the muscle (not including the thickness of fascial muscle layers).
Change in IOTF | Measured for 5 breaths in the 30 minutes for each training block (A1-4 & B1-4; cumulative 4hours)
  Internal oblique muscle thickening fraction, calculated as (internal oblique muscle thickness at end-inspiration - internal oblique muscle thickness at end-expiration) / internal oblique muscle thickness at end-expiration [dimensionless]. Muscle thickness will be measured in millimeters using M-mode ultrasound with the probe placed perpendicular to the muscle (not including the thickness of fascial muscle layers).
Change in MIP (cmH2O) | Measured during an expiratory hold of ≤ 30 seconds between each training block (AH0-4 & BH0-4; cumulative ≤ 5 minutes)
  Maximal inspiratory pressure
Change in MEP (cmH2O) | Measured during an inspiratory hold of ≤ 30 seconds between each training block (AH0-4 & BH0-4; cumulative ≤ 5 minutes)
  Maximal expiratory pressure
Change in ∆Pocc (cmH2O) | Measured during an expiratory hold of ≤ 30 seconds between each training block (AH0-4 & BH0-4; cumulative ≤ 5 minutes)
  Airway occlusion pressure
Change in NVE (ml/µv) | Measured at each breath during 30 minutes for each training block (A1-4 & B1-4; cumulative 4hours)
  Neuroventilatory efficiency, calculated as tidal volume divided by delta Edi. It is measured at a pressure support of 7 cmH2O, i.e. NOT during a zero assist manoeuvre.
Change in TV (ml) | Measured at each breath during 30 minutes for each training block (A1-4 & B1-4; cumulative 4hours)
  Tidal volume
Change in ∆Edi (µV) | Measured at each breath during 30 minutes for each training block (A1-4 & B1-4; cumulative 4hours)
  Increase in electrical activity of the diaphragm (Edi) during inspiration, calculated as Edi high - Edi low.
Change in Pplat (cmH2O) | Measured at each breath during 30 minutes for each training block (A1-4 & B1-4; cumulative 4hours)
  Airway plateau pressure
Change in static PEEP (cmH2O) | Measured during an expiratory hold of ≤ 30 seconds between each training block (AH0-4 & BH0-4; cumulative ≤ 5 minutes)
  Postive end-expiratory pressure as measured during an expiratory hold.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe G Jorens, MD, PhD, Principal Investigator — Head of the department of critical care medicine, Antwerp University Hospital
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Time series of NVE-ZAM will be plotted per participant and reported in a publication.